CLINICAL TRIAL: NCT05875870
Title: Effects of Bright-light Exposure Combined With Specific Exercise Training (BEST) Program on Sleep-Wake Rhythm, Physical and Psychological Symptoms, and Quality of Life of Patients With Thoracic Cancer: A Series Study.
Brief Title: Effects of Bright-light Exposure Combined With Specific Exercise Training (BEST) Program in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-04-003B
Record Dates: First submitted 2023-05-01; First posted 2023-05-25 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Lung Neoplasm; Esophageal Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The rehabilitation program is composed of two parts: six-week bright-light exposure program and an exercise program.
  Interventions: Behavioral: Daylight exposure combine walking
- Active control group (Active Comparator): The active control group receives six weeks of a stretching exercise.
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Daylight exposure combine walking — 1. Out-door of bright-light exposure in the morning (36 min/day, 7 times/week) for six weeks.
  2. Tailored to the individual patient with moderate intensity of walking (3 sessions/week) for six weeks. Duration of each session depends on one-on-one exercise consultation via communication software (LINE App). The duration of walking in week 1 is 15 minutes, then increasing 5 minutes each week if the patient has tolerance. If the patient cannot tolerate the duration, the coach will instruct to keep the same duration for the following week. Basically, the goal of duration in week six is 40 minutes.
  3. Weekly exercise consultation via communication software (LINE App).
  4. Teaching strategy includes one-on one instruction (hard-copy of teaching manual), video, and webpage.
  Arms: Experimental group
Behavioral: Stretching exercise — The stretching exercise includes two movements for the upper body and two movements for the lower body, 10 minutes each time, three times a week, for 6 weeks.
  The researcher will explain to the participants about how to perform the stretching exercise, according to an instruction manual (hardcopy) for the exercise regimen.
  A video is shown to the participants (the content same as hardcopy of education manual).
  Arms: Active control group

SUMMARY:
This study plans to investigate the effectiveness of six-week light exposure combined with an exercise training program on improving sleep-wake rhythm, physical and mental symptoms, quality of life, one-year recurrence rate, and one-year survival rate of patients with lung and esophageal cancer.

DETAILED DESCRIPTION:
This study plans to investigate the effectiveness of six-week light exposure combined with an exercise training program on improving sleep-wake rhythm, physical and mental symptoms, quality of life, one-year recurrence rate, and one-year survival rate of patients with lung and esophageal cancer.

Two groups, parallel, randomly assigned clinical trials, long-term follow-up, repeated measurement (pre-test, 6th week, 12th week, 6th month, 12th month, five times in total), and a design of single center recruitment. The experimental group receiving an intervention comprised six weeks of light exposure combined with exercise training. The active control group receiving six weeks of stretching exercise. With a double-blind study design of participant blind and outcomes assessor blind, subjects were recruited from the thoracic surgery clinic and thoracic surgery ward of a medical center in northern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed primary lung cancer or esophageal cancer, from the first stage to the third stage.
2. At least 20 years of age.
3. Able to communicate in Mandarin Chinese or Taiwanese.
4. Literate and free from cognitive disabilities.
5. The attending physician agrees to participate in the study.
6. Those who can connect to the Internet with mobile devices such as computers, mobile phones, and tablets, or those whose family members can assist in the operation.
7. Those with Karnofsky Performance Scale (KPS) greater than or equal to 70 points.
8. Those who are hospitalized for lung cancer or esophageal cancer lesion resection.

Exclusion Criteria:

1. Congestive heart failure.
2. Orthopedic diseases of the lower extremities that limit one's walking ability.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Sleep-wake rhythm | Baseline
  Using Actigraph to measure sleep-wake rhythm. The parameter including 24-h correlation coefficient(r24), in bed less than out of bed dichotomy index (I < O), midline estimating statistic of rhythm (MESOR), and amplitude…etc.
Sleep-wake rhythm | Change from baseline sleep-wake rhythm at 6th week
  Using Actigraph to measure sleep-wake rhythm. The parameter including 24-h correlation coefficient(r24), in bed less than out of bed dichotomy index (I < O), midline estimating statistic of rhythm (MESOR), and amplitude…etc.
Sleep-wake rhythm | Change from baseline sleep-wake rhythm at 12th week
  Using Actigraph to measure sleep-wake rhythm. The parameter including 24-h correlation coefficient(r24), in bed less than out of bed dichotomy index (I < O), midline estimating statistic of rhythm (MESOR), and amplitude…etc.
Sleep-wake rhythm | Change from baseline sleep-wake rhythm at 6th month
  Using Actigraph to measure sleep-wake rhythm. The parameter including 24-h correlation coefficient(r24), in bed less than out of bed dichotomy index (I < O), midline estimating statistic of rhythm (MESOR), and amplitude…etc.
Sleep-wake rhythm | Change from baseline sleep-wake rhythm at 12th month
  Using Actigraph to measure sleep-wake rhythm. The parameter including 24-h correlation coefficient(r24), in bed less than out of bed dichotomy index (I < O), midline estimating statistic of rhythm (MESOR), and amplitude…etc.

SECONDARY OUTCOMES:
Subjective sleep quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Subjective sleep quality (Pittsburgh Sleep Quality Index, PSQI) | Change from baseline sleep-wake rhythm at 6th week
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Subjective sleep quality (Pittsburgh Sleep Quality Index, PSQI) | Change from baseline sleep-wake rhythm at 12th week
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Subjective sleep quality (Pittsburgh Sleep Quality Index, PSQI) | Change from baseline sleep-wake rhythm at 6th month
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Subjective sleep quality (Pittsburgh Sleep Quality Index, PSQI) | Change from baseline sleep-wake rhythm at 12th month
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Objective sleep quality: total sleep time | Baseline
  Using actigraph to measure total sleep time (min/night)
Objective sleep quality: total sleep time | Change from baseline total sleep time at 6th week
  Using actigraph to measure total sleep time (min/night)
Objective sleep quality: total sleep time | Change from baseline total sleep time at 12th week
  Using actigraph to measure total sleep time (min/night)
Objective sleep quality: total sleep time | Change from baseline total sleep time at 6th month
  Using actigraph to measure total sleep time (min/night)
Objective sleep quality: total sleep time | Change from baseline total sleep time at 12th month
  Using actigraph to measure total sleep time (min/night)
Objective sleep quality: sleep onset latency | Baseline
  Using actigraph to measure sleep onset latency (min/night)
Objective sleep quality: sleep onset latency | Change from baseline sleep onset latency at 6th week
  Using actigraph to measure sleep onset latency (min/night)
Objective sleep quality: sleep onset latency | Change from baseline sleep onset latency at 12th week
  Using actigraph to measure sleep onset latency (min/night)
Objective sleep quality: sleep onset latency | Change from baseline sleep onset latency at 6th month
  Using actigraph to measure sleep onset latency (min/night)
Objective sleep quality: sleep onset latency | Change from baseline sleep onset latency at 12th month
  Using actigraph to measure sleep onset latency (min/night)
Objective sleep quality: sleep efficiency | Baseline
  Using actigraph to measure sleep efficiency (percentage)
Objective sleep quality: sleep efficiency | Change from baseline sleep efficiency at 6th week
  Using actigraph to measure sleep efficiency (percentage)
Objective sleep quality: sleep efficiency | Change from baseline sleep efficiency at 12th week
  Using actigraph to measure sleep efficiency (percentage)
Objective sleep quality: sleep efficiency | Change from baseline sleep efficiency at 6th month
  Using actigraph to measure sleep efficiency (percentage)
Objective sleep quality: sleep efficiency | Change from baseline sleep efficiency at 12th month
  Using actigraph to measure sleep efficiency (percentage)
Objective sleep quality: wake after sleep onset | Baseline
  Using actigraph to measure wake after sleep onset (min/night)
Objective sleep quality: wake after sleep onset | Change from baseline wake after sleep onset at 6th week
  Using actigraph to measure wake after sleep onset (min/night)
Objective sleep quality: wake after sleep onset | Change from baseline wake after sleep onset at 12th week
  Using actigraph to measure wake after sleep onset (min/night)
Objective sleep quality: wake after sleep onset | Change from baseline wake after sleep onset at 6th month
  Using actigraph to measure wake after sleep onset (min/night)
Objective sleep quality: wake after sleep onset | Change from baseline wake after sleep onset at 12th month
  Using actigraph to measure wake after sleep onset (min/night)
Anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Baseline
  The scale consists of seven items each for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) was scored on a 4-point scale from 0 (not at all) to 3 (very much so). Higher scores indicated higher anxiety or depression levels.
Anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Change from baseline anxiety and depression at 6th week
  The scale consists of seven items each for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) was scored on a 4-point scale from 0 (not at all) to 3 (very much so). Higher scores indicated higher anxiety or depression levels.
Anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Change from baseline anxiety and depression at 12th week
  The scale consists of seven items each for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) was scored on a 4-point scale from 0 (not at all) to 3 (very much so). Higher scores indicated higher anxiety or depression levels.
Anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Change from baseline anxiety and depression at 6th month
  The scale consists of seven items each for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) was scored on a 4-point scale from 0 (not at all) to 3 (very much so). Higher scores indicated higher anxiety or depression levels.
Anxiety and depression (Hospital Anxiety and Depression Scale, HADS) | Change from baseline anxiety and depression at 12th month
  The scale consists of seven items each for anxiety and depression. Each item of the anxiety subscale (HADS-A) and the depression subscale (HADS-D) was scored on a 4-point scale from 0 (not at all) to 3 (very much so). Higher scores indicated higher anxiety or depression levels.
Quality of life (European Organization for Research and Treatment of cancer quality of life questionnaire) | Baseline
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life (European Organization for Research and Treatment of cancer quality of life questionnaire) | Change from baseline quality of life at 6th week
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life (European Organization for Research and Treatment of cancer quality of life questionnaire) | Change from baseline quality of life at 12th week
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life (European Organization for Research and Treatment of cancer quality of life questionnaire) | Change from baseline quality of life at 6th month
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life (European Organization for Research and Treatment of cancer quality of life questionnaire) | Change from baseline quality of life at 12th month
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Recurrent rate | 12th month after recruitment
  Chart review to determine whether cancer has recurred for participant one year after diagnosis.
Survival rate | 12th month after recruitment
  Chart review to determine whether participant survived one year after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taipei Veterans General Hospital, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Result] Chen HM, Cheung DST, Lin YY, Wu YC, Liu CY, Lin KC, Lin YJ, Lin CC. Relationships of exercise timing with sleep, fatigue and rest-activity rhythms of lung cancer patients in Taiwan: An exploratory study. Eur J Cancer Care (Engl). 2020 Jul;29(4):e13233. doi: 10.1111/ecc.13233. Epub 2020 Feb 25. PMID 32100388
- [Result] Chen HM, Lee MC, Tian JY, Dai MF, Wu YC, Huang CS, Hsu PK, Duong LT. Relationships Among Physical Activity, Daylight Exposure, and Rest-Activity Circadian Rhythm in Patients With Esophageal and Gastric Cancer: An Exploratory Study. Cancer Nurs. 2024 Mar-Apr 01;47(2):112-120. doi: 10.1097/NCC.0000000000001188. Epub 2023 Jan 14. PMID 36728167
- [Result] Chen HM, Lin YY, Wu YC, Huang CS, Hsu PK, Chien LI, Lin YJ, Huang HL. Effects of Rehabilitation Program on Quality of Life, Sleep, Rest-Activity Rhythms, Anxiety, and Depression of Patients With Esophageal Cancer: A Pilot Randomized Controlled Trial. Cancer Nurs. 2022 Mar-Apr 01;45(2):E582-E593. doi: 10.1097/NCC.0000000000000953. PMID 33813524
- [Result] Chen HM, Tsai CM, Wu YC, Lin KC, Lin CC. Randomised controlled trial on the effectiveness of home-based walking exercise on anxiety, depression and cancer-related symptoms in patients with lung cancer. Br J Cancer. 2015 Feb 3;112(3):438-45. doi: 10.1038/bjc.2014.612. Epub 2014 Dec 9. PMID 25490525
- [Result] Chen HM, Tsai CM, Wu YC, Lin KC, Lin CC. Effect of walking on circadian rhythms and sleep quality of patients with lung cancer: a randomised controlled trial. Br J Cancer. 2016 Nov 22;115(11):1304-1312. doi: 10.1038/bjc.2016.356. Epub 2016 Nov 3. PMID 27811855
- [Result] Chen HM, Wu YC, Tsai CM, Tzeng JI, Lin CC. Relationships of Circadian Rhythms and Physical Activity With Objective Sleep Parameters in Lung Cancer Patients. Cancer Nurs. 2015 May-Jun;38(3):215-23. doi: 10.1097/NCC.0000000000000163. PMID 24945266
- See also: Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable — https://pubmed.ncbi.nlm.nih.gov/31626055/